CLINICAL TRIAL: NCT03398954
Title: Screening Out Rate and Clinical Management of Familial Hypercholesterolemia： a Prospective Pilot Study in China Outpatient Department
Brief Title: a Prospective Pilot Study of Screening Out Rate and Clinical Management of Familial Hypercholesterolemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Cardiovascular Association (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20177276
Record Dates: First submitted 2017-12-20; First posted 2018-01-16 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-01

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Primary Objective To estimate the prevalence of clinical diagnosed familial hypercholesterolemia, as well as the clinical characteristics and current treatment, with applying China recent issued FH screening protocol in pilot outpatient department of China.
2. Study Design The study is a prospective observational research study of clinical diagnoses FH patients in outpatient department in pilot hospitals to evaluate the screening out rate and the clinical feature and management of FH patients including HoFH, with applying China recent issued FH screening protocol.
3. Eligibility 3.1.Inclusion Criteria Written inform consent provided. Male and female cardiovascular outpatients and inpatients with LDL-C>4.65mmol/L if statin naïve or LDL-C>3.7mmol/L if on statin treatment before enrollment during Sept.2017 to Sept. 2019.

   3.2Exclusion Criteria Subjects who cannot understand study procedure Subjects diagnosed as secondary dyslipidemia
4. Primary Endpoint

   * The screening out rate of clinical diagnosed familial hypercholesterolemia, with applying China recent issued FH screening protocol in subjects with LDL-C>4.65mmol/L if statin naïve or LDL-C>3.7mmol/L if on statin treatment in pilot outpatient department of China.
   * The clinical characteristics of clinical diagnosed FH patients(including HoFH and HeFH), including: demography, medical history, family history, sign and symptoms, lab testing and cardiovascular imagine result.
   * The pharmaceutical therapy for clinical diagnosed FH patients (including HoFH and HeFH), including the type of medication, proportion for each medication, dosage and treatment duration.

DETAILED DESCRIPTION:
1. Objective 1.1.Primary Objective To estimate the prevalence of clinical diagnosed familial hypercholesterolemia, as well as the clinical characteristics and current treatment, with applying China recent issued FH screening protocol in pilot outpatient department of China.

   1.2.Secondary Objective To describe parameters related to clinical management of diagnosed FH, including patient demographics and characteristics, LDL-C and triglyceride concentrations, use of lipid modifying therapies, and outcomes over time.

   1.3.Exploratory To describe how China FH screening protocol fits in the practice when compared with DLCN.

   To explore the multi-disciplinary practical pattern of FH patient management
2. Endpoint(s)/Outcome(s) Assessment 2.1.Endpoint(s) 2.1.1.Primary Endpoint The screening out rate of clinical diagnosed familial hypercholesterolemia, with applying China recent issued FH screening protocol in subjects with LDL-C>4.65mmol/L if statin naïve or LDL-C>3.7mmol/L if on statin treatment in pilot outpatient department of China.

   The clinical characteristics of clinical diagnosed FH patients(including HoFH and HeFH), including: demography, medical history, family history, sign and symptoms, lab testing and cardiovascular imagine result.

   The pharmaceutical therapy for clinical diagnosed FH patients (including HoFH and HeFH), including the type of medication, proportion for each medication, dosage and treatment duration.

   2.1.2.Secondary Endpoint LDL-C level during the follow up period The pharmaceutical therapy for clinical diagnosed FH patients (including HoFH and HeFH), including the type of medication, proportion for each medication, dosage and treatment duration during the follow up period.

   Achievement of 2016 China guideline defined target LDL-C levels; <2.6mmol/L (high risk), <1.8mmol/L (very high risk) Incidence of cardiovascular event (CV death, all-cause mortality, non-fatal MI, non-fatal stroke).

   2.1.3Exploratory Endpoint The difference of FH screening out rate between China criteria and DLCN. 2.2.Study Parameters 2.2.1.Baseline Data Collection Demography data:Age,Gender, Personal history:Premature CHD history of the subject (male: <55yrs, female: <65yrs),Premature PAD or cerebral vascular disease of the subject (male: <55yrs, female: <65yrs),Smoking, Medical history:PAD,DM,Hypertension,Heart Failure,Stroke,MI,CABG/PTCA/PCI,CKD Family history:Premature CHD within 2nd grade relatives (1st grade relatives, male: <55yrs, female: <60yrs; 2nd grade relatives, male: <50yrs, female: <55yrs),FH diagnosis within 2nd grade relatives Physical exam:Height,Weight,BMI,Corneal Arcus,Xanthoma,Achilles tender thickness Lab:LDL-C,HDL-C ,TC,TG,Lp(a),ALT,AST,CK,Glucose,Creatinine,Urea nitrogen,Inflammatory biomarker, including hs CRP ECG Cardiovascular imagine:CAG(optional),Myocardial radionuclide imaging (optional),UCG(annually),Carotid plaques measure(annually) Lipid modification therapy:Statin(type, dosage),Non-Statin(type, dosage) Apheresis 2.2.2Study Follow Up Period Data Collection Lab:LDL-C,HDL-C,TC,TG,Lp(a),ALT,AST,CK,Glucose,Creatinine,Urea nitrogen Inflammatory biomarker, including hs CRP Cardiovascular imagine:CAG(optional),Myocardial radionuclide imaging (optional),UCG(annually),Carotid plaques(annually) Lipid modification therapy:Statin(type, dosage),Non-Statin(type, dosage) Apheresis; Achievement of 2016 China guideline defined target LDL-C levels; <2.6mmol/L (high risk), <1.8mmol/L (very high risk); Incidence of cardiovascular event (CV death, all-cause mortality, non-fatal MI, non-fatal stroke).
3. STATISTICAL ANALYSIS 3.1.Statistical Inference No formal hypothesis will be tested in this study. This study will estimate the prevalence of Familial Hypercholesterolemia and the related 95% confidence interval in the China outpatient population in pilot hospitals.

   3.2.Sample Size Considerations Based on initial feasibility analyses,revealed an approximate annual patient population in cardiology outpatients is 1,000pts/month(50pts/day*20days) with lipid profile measured to be screened. It is estimated that about 3000 patients out of cardiology department will measure their lipid profile in the clinical laboratory, the working days for the outpatient department is defined as 10mon, then total patients number in the outpatient will be about 4000pts/mon/center*10mon=40,000/center/yr. The prevalence of suspected patients based on LDL-C level is 0.47%, then 188 clinical diagnosed patients/center/year to be transited to the follow up period. Based on the planned site number of 6, total patient to be enrolled to this study will be 1128. Based on the prevalence of HoFH is near 1/160,000~1/300,000, it is estimated that 1~2 HoFH patients will be identified from this patient population.

   3.3.Planned Analyses All summaries of the data will be descriptive in nature. For categorical variables (including the primary outcome measure), the frequency and percentage, with 95% confidence interval, will be given. Summary statistics for continuous variables will include the number of subjects, mean, median, standard deviation or standard error, 25th percentile (Q1), 75th percentile (Q3), minimum, and maximum. The outcomes over time data will be evaluated using time to event analyses/Cox proportional hazards models. All planned analyses will be descriptive. SAS version 9.2 (or a newer version) will be used for all Data Management and Statistical Analyses.

   3.3.1.Description of Study Enrollment All subjects enrolled into the study who meet the inclusion criteria will be included in the full analysis set and will be included in all summaries and analyses.

   3.3.2.Description of Subject/Patient Characteristics Clinical characteristics of subjects in the study will be summarized. Measurements such as age will be based on the status at the start of the observation period for the subject, and clinical characteristics such as CV events will be captured throughout the 3.3.3.Primary Analysis Primary Objective

   -To estimate the screen out rate of clinical diagnosed familial hypercholesterolemia in outpatient department of China.

   Prevalence: Prevalence of suspected FH will be estimated using the patients' data who visited the outpatients department in pilot hospitals and with measurable LDL-C data and validated by China criteria and DNCL respectively. Prevalence will be reported annually for the years 2017-2019.

   -To describe parameters related to clinical management of diagnosed FH, including patient demographics and characteristics, LDL-C and triglyceride concentrations, use of lipid modifying therapies, and outcomes over time.

   Patient demographics: Analyses of prevalence will be estimated for the following demographic characteristics: age, gender, and region.

   Patient clinical characteristics: The proportion of patients, calculated as percentage of patients, for each of the following: BMI (obese/not obese), diabetes, CKD, hypertension, any CVD history / number of CV events, smoking status (current / previous). These will be measured both at baseline (time of FH diagnosis).

   Current use of lipid-modifying therapies over time: Proportion of patients using LMT. Analyses by type, dose and frequency will analysis with description statistical method.

   Secondary Objective
   * LDL-C concentrations over time. The LDL-C level will be follow up to the end of study.
   * Use of lipid-modifying therapies over time。 Proportion of patients using LMT. Analyses by type, dose and frequency, and the proportion of patients on a high-intensity statin regime and with high LDL-C will be performed.
   * Proportion of patients within and at distance from 2016 China guideline's LDL-C target.

   This will be calculated as the percentage of patients within 2016 China guideline LDL-C target (<2.6 mmol/L, <1.8 mmol/L). LDL-C measurements will be followed up to the end of study.

   -Incidence of fatal and non-fatal cardiovascular events The proportion of patients having a fatal or non-fatal cardiovascular event will be calculated. Since there may be competing risks with fatal / non-fatal events, analyses will be performed separately, and in combination. All events occurring from date of enrollment of the study onwards will be included.

   3.3.4.General Considerations The first primary objective and all secondary objectives will be addressed through descriptive statistics. The CV outcome will be evaluated using time to event analyses.

   3.3.5.Missing or Incomplete Data and Lost to Follow-up There are two types of data in this study. For different data types, we will apply different methods to handle missing data.

   For Medical records abstraction:

   The missing age values will be imputed as the overall median to avoid case-wise deletions. For some of the patients, certain physiological indicators were not measured during hospitalization. These variables will be treated as a specific "unmeasured" subgroup with clinical significance because not measured is not equal to "missing" and may influence the outcomes. If we fit these variables as continuous in the models, we could only arbitrarily consider these "unmeasured" as missing value as inappropriate. Imputation also has limitations. Thus, to keep the models consistent with the features of data, we will transform certain continuous variables into categorical ones, created dummy variables accordingly, and including a specific category to indicate unmeasured.

   For Baseline and follow-up questionnaires:

   Site investigators completed the questionnaires in an electronic data capture program on a tablet computer (which allows real-time logic checks to ensure the accuracy and completeness of data). All questions were required to be answered, except those that were not applicable. There were options of "refuse to answer" and "don't know" for each question.
4. SAFETY DATA COLLECTION, RECORDING, AND REPORTING Due to the non-interventional nature of this study, no pro-active safety data collection will take place. Only spontaneously mentioned safety events and in-hospital clinical events will be collected in this study, and reported follow by local regulation.

ELIGIBILITY:
Inclusion Criteria:

* Written inform consent provided.
* Male and female cardiovascular outpatients and inpatients with LDL-C>4.65mmol/L if statin naïve or LDL-C>3.7mmol/L if on statin treatment before enrollment during Sept.2017 to Sept. 2019.

Exclusion Criteria:

* Subjects who cannot understand study procedure
* Subjects diagnosed as secondary dyslipidemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the primary objective the study population will comprise all patients with a documented LDL-C>4.65mmol/L if statin naïve and LDL-C>3.7mmol/L if on statin treatment before enrollment in the outpatient department of pilot hospitals from Sept. 2017-Sept. 2019.
Sampling Method: Probability Sample
Enrollment: 1128 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The screening out rate of FH | 2 years
  The screening out rate of clinical diagnosed familial hypercholesterolemia, with applying China recent issued FH screening protocol in subjects with LDL-C>4.65mmol/L if statin naïve or LDL-C>3.7mmol/L if on statin treatment in pilot outpatient department of China.
The clinical characteristics of clinical diagnosed FH patients | 2 years
  The clinical characteristics of clinical diagnosed FH patients(including HoFH and HeFH), including: demography, medical history, family history, sign and symptoms, lab testing and cardiovascular imagine result
The pharmaceutical therapy for clinical diagnosed FH patients | 2 years
  The pharmaceutical therapy for clinical diagnosed FH patients (including HoFH and HeFH), including the type of medication, proportion for each medication, dosage and treatment duration

SECONDARY OUTCOMES:
LDL-C concentrations over time | 2 years
  LDL-C level during the follow up period
Use of lipid-modifying therapies over time | 2 years
  The pharmaceutical therapy for clinical diagnosed FH patients (including HoFH and HeFH), including the type of medication, proportion for each medication, dosage and treatment duration during the follow up period
Proportion of patients within and at distance from 2016 China guideline's LDL-C target | 2 years
  Achievement of 2016 China guideline defined target LDL-C levels; <2.6mmol/L (high risk), <1.8mmol/L (very high risk)
Incidence of cardiovascular event | 2 years
  Incidence of cardiovascular event (CV death, all-cause mortality, non-fatal MI, non-fatal stroke)

CONTACTS AND LOCATIONS:
Overall Officials: huo yong, master, Principal Investigator — Peking University First Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qureshi N, Da Silva MLR, Abdul-Hamid H, Weng SF, Kai J, Leonardi-Bee J. Strategies for screening for familial hypercholesterolaemia in primary care and other community settings. Cochrane Database Syst Rev. 2021 Oct 7;10(10):CD012985. doi: 10.1002/14651858.CD012985.pub2. PMID 34617591